CLINICAL TRIAL: NCT01916434
Title: FIsh for a Sustainable Healthy Diet In Scottish Households Study
Brief Title: Farmed Fish Human Intervention Study
Acronym: FISHDISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2005
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Disease
Keywords: Farmed fish; Dietary intervention; Long-term intervention; Omega-3 index; Cardiovascular risk markers; Coagulation and endothelial activation; Bleeding time; Inflammation; Oxidative stress; Gut health; Micronutrient availability
MeSH Terms: conditions — Cardiovascular Diseases; Thrombosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Pufa Salmon Fillets (Experimental): High EPA/DHA levels in feed and in salmon fillets (~15% of total feed fatty acids, equal to wild salmon), 2 salmon fillets per week for 18 weeks, on top of habitual fish consumption.
  Interventions: Other: High PUFA Salmon Fillets
- Sustainable PUFA salmon (Experimental): 'Sustainable' levels of EPA/DHA in feed and in salmon fillets (~6-8% of total feed fatty acids), 2 salmon fillets per week for 18 weeks, on top of habitual fish consumption
  Interventions: Other: Sustainable PUFA salmon
- No salmon (Placebo Comparator): The placebo group will continue to consume their habitual diet
  Interventions: Other: No salmon

INTERVENTIONS:
Other: High PUFA Salmon Fillets — High EPA/DHA levels in feed and in salmon fillets (~15% of total feed fatty acids, equal to wild salmon), 2 salmon fillets per week for 18 weeks, on top of habitual fish consumption.
  Arms: High Pufa Salmon Fillets
Other: Sustainable PUFA salmon — 'Sustainable' levels of EPA/DHA in feed and in salmon fillets (~6-8% of total feed fatty acids), 2 salmon fillets per week for 18 weeks, on top of habitual fish consumption.
  Arms: Sustainable PUFA salmon
Other: No salmon — The placebo group will continue to consume their habitual diet.
  Arms: No salmon

SUMMARY:
Consumption of fish can help to prevent cardiovascular disease. The precise way in which fish is beneficial is not fully understood. This is important to find out as fish consists of a complex mixture of fatty acids and micronutrients such as vitamin D and selenium that could individually, or collectively, be responsible for the beneficial effects.

Fish farming in Scotland is playing an increasingly important role in the provision of fish for human consumption. But issues with sustainability of raw materials are requiring fish farming to reformulate fish diets, which may affect the levels of beneficial omega-3 fatty acids and other components in fish.

In this study we will be comparing the long-term health effects of eating two portions a week of Scottish salmon raised on a traditional fish diet versus eating two portions a week of Scottish salmon raised on a more sustainable fish diet. In addition, we will be looking at differences in health outcomes when eating two portions a week of either Scottish salmon, compared with eating no fish at all.

DETAILED DESCRIPTION:
Aquaculture has the potential to take the pressure off wild fish stocks whilst meeting the dietary needs of the population for omega 3 fatty acids and other key nutrients such as vitamin D. The industry is working hard to improve sustainability - between 1995 and 2006 it has been estimated that the input to output ratios for salmon improved from 7.5 to 4.9 and trout from 6.0 to 3.4- but there is a need to do more. Reductions in fish stocks and catch quotas, in addition to sustainability considerations, mean that farmed fish may have to be raised on vegetable oils for example but this may reduce the omega 3 content and may affect the content of other nutrients. Fish are an important component of the diet and there is a need to understand the effect of pressures from sustainability on methods of production and the health giving properties of fish. We have now been commissioned by the Scottish Government's Rural and Environment Science and Analytical Services Division (RESAS) to do research on the health effects of Scottish farmed fish fed different feeding regimes in the Scottish population, and assess how differential effects in measured health outcomes could be related to fish composition.

Consumption of fish or omega-3- fatty acids from fish reduces coronary heart disease mortality, the leading cause of death in developed nations. The precise way in which fish provides benefit is not fully understood. This is important as fish and fish oils consist of a complex mixture of fatty acids and micronutrients that could individually, or collectively, be responsible for the beneficial effects. Aquaculture in Scotland is playing an increasingly important role in the provision of fish for human consumption, but issues with sustainability are requiring aquaculture to replace traditional fish oil and meal in formulated fish diets by oil from more sustainable sources, which may affect the levels of beneficial omega-3 fatty acids (EPA and DHA) and other components in fish. We will investigate the health effects of consuming two portions oily fish (Scottish farmed salmon) per week (current UK recommendation) using fish raised on different feeding regimes.

HYPOTHESIS

The health effects of consuming two portions oily fish (Scottish farmed salmon) per week (current UK recommendation) will be different for fish raised on different feeding regimes, primarily in terms of improving the omega-3 index.

OBJECTIVE

The main objective of this proposed study is to determine 1) whether the health benefits of consuming two portions of Scottish farmed salmon per week that have been fed a diet high in fish oil and fish meal significantly outweigh the health benefits of consuming two portions of Scottish farmed salmon per week that have been fed a diet with more sustainable levels of fish meal and fish oil, and 2) whether the difference in health benefits could justify the use of less sustainable dietary regimes for farmed fish.

ELIGIBILITY:
Inclusion criteria: Healthy men and women aged 35-75 years BMI ranging from 18-35 kg/m2 Blood pressure below 160/90 mmHg; Total cholesterol < 8.00 mmol/L Total/HDL cholesterol < 6 mmol/L Fasting plasma glucose , 7 mmol/L Having a 10-20% risk for developing cardiovascular disease within the next 10 years based on the ASSIGN calculation (http://cvrisk.mvm.ed.ac.uk/index.htm) including the following factors: age, gender, number of cigarettes smoked per day, Scottish Index of Multiple Deprivation (SIMD)/postcode, systolic blood pressure, levels of total and HDL cholesterol and family history of cardiovascular disease, or having at least one additional risk factor such as being over 50 years old, BMI above 25 kg/m2, elevated triglyceride levels (> 1.7 mmol/L) or elevated glucose levels (> 5.6 mmol/L); platelet count > 1709/L haematocrit above 40 % for males and above 35 % for females haemoglobin above 130 g/L for males and above 115 g/L for females

Exclusion criteria Regularly taking aspirin or aspirin-containing drugs, or other anti-inflammatory drugs; Taking drugs or herbal medicines known to alter the haemostatic system in general; Taking any medicine known to affect lipid metabolism; Taking certain dietary supplements/multivitamin tablets; Diagnosis of diabetes, hypertension, renal, hepatic, haematological disease or coronary heart disease; Unsuitable veins for blood sampling; Inability to understand the participant information sheet; inability to speak, read and understand the English language.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the omega-3 index | At baseline and after 18 weeks salmon consumption
  The Omega-3 index will be measured by GC-MS. An optimal target level of the Omega-3 Index is 8%, and an undesirable level is less than 4%, with 4-8% being an intermediate-risk zone.

SECONDARY OUTCOMES:
Change in cardiovascular risk markers | At baseline, after 9 weeks and after 18 weeks salmon consumption
  This study will include the measurement of standard risk markers of cardiovascular disease at the start, middle and end of the intervention period, including lipoprotein metabolism (total cholesterol, LDL cholesterol, HDL cholesterol) and metabolic markers (glucose, insulin, triglycerides and non-esterified fatty acids to calculate HOMA-IR and revised QUICKI). We will also measure 24-hrs ambulatory blood pressure.

OTHER OUTCOMES:
Bleeding time as measured by the platelet function analyzer (PFA-100) | At baseline and after 18 weeks salmon consumption
  The PFA-100 simulates high shear platelet function in citrated blood within disposable test cartridges with membranes coated with either collagen/epinephrine (CEPI) or collagen/ADP (CADP). The presence of these platelet activators and the high shear rates under the standardised conditions result in platelet adhesion, activation and aggregation resulting in formation of a platelet plug within the aperture. Platelet function is thus measured as a function of the time it takes to occlude the aperture.
Markers of coagulation and endothelial activation. | At baseline and after 18 weeks salmon consumption
  Fibrinogen is a principle plasma glycoprotein involved in blood clotting. Plasma clottable fibrinogen levels will be measured by Clauss method on a semi-automated coagulometer using Fibrinogen assay thrombin reagent from Helena Biosciences, England. Von Willebrand factor (vWF) is another plasma glycoprotein involved in coagulation and an established marker of endothelial activation or damage. Plasma levels of vWF will be measured by an in-house ELISA using polyclonal antibodies and horseradish peroxidase-conjugated antibody from DAKO Ltd, Denmark. P-selectin is a cell adhesion molecule present in platelet granules and (to a lesser extent) in endothelial cells. sP-selectin levels in fasted blood plasma will be measured in duplicate by ELISA (Bender Med Systems)
Markers of inflammation. | At baseline and after 18 weeks salmon consumption
  CRP is an acute phase protein synthesised by the liver in response to inflammatory stimuli, especially the cytokine IL-6. hsCRP will be measured in duplicate by an ultra sensitive, double antibody ELISA. Soluble -ICAM is a marker of endothelial activation and inflammation, during which it promotes leucocyte adherence to the endothelium. Plasma soluble I-CAM levels will be measured in duplicate by ELISA (Bender Med Systems). Epoxyeicosatrieonic acids (EETs) are anti-inflammatory and cardioprotective compounds. Their availability and metabolism are regulated by the enzyme soluble epoxide hydrolase (sEH), which in turn is affected by EPA. EETs will be measured in platelets using LC-MS/MS.
Markers of oxidative stress. | At baseline and after 18 weeks salmon consumption
  F2-isoprostanes are currently considered as reference biomarkers for lipid peroxidation and will be measured by LC-MS/MS.
Markers of micronutrient availability | At baseline and after 18 weeks salmon consumption
  Selenium in incorporated into proteins within the body, many of which are antioxidants that protect the body against oxidative damage. Selenium is transported across the body within the protein, selenoprotein P (SEPP-1). Selenium status will be measured by assaying plasma selenium levels (by ICP-MS) and by quantification of plasma SEPP-1 levels (by an in-house ELISA). Iodine status will be measured by assaying urinary iodine levels (by ICP-MS) and vitamin D status will be assessed by measuring plasma 25-hydroxy vitamin D (using HPLC and LC/MS/MS).
Markers of gut health | At baseline and after 18 weeks salmon consumption
  Faecal samples will be collected for the isolation of faecal waters to measure NFkb activation, micronutrient levels, genetic health and antioxidant potential (ORAC, TRAC etc), as well as the measurement of stool content and stool pH.
Markers of genetic health | At baseline and after 18 weeks salmon consumption
  The buffy coat from spun whole blood samples will be collected to measure patterns of DNA methylation contributing to epigenetic inheritance.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje De Roos, Msc, PhD, Principal Investigator — University of Aberdeen Rowett Institute of Nutrition and Health
Locations (1):
- Rowett Institute of Nutrition and Health, Human Nutrition Unit, Aberdeen, United Kingdom

REFERENCES:
- [Derived] de Roos B, Wood S, Bremner D, Bashir S, Betancor MB, Fraser WD, Duthie SJ, Horgan GW, Sneddon AA. The nutritional and cardiovascular health benefits of rapeseed oil-fed farmed salmon in humans are not decreased compared with those of traditionally farmed salmon: a randomized controlled trial. Eur J Nutr. 2021 Jun;60(4):2063-2075. doi: 10.1007/s00394-020-02396-w. Epub 2020 Oct 5. PMID 33015732